CLINICAL TRIAL: NCT04941677
Title: Exploration of the Relationships Between Vocational Performances Ans Sensorimotor Factors of Hands in Schizophrenia
Brief Title: Exploring Hand Function in People With Schizophrenia Based on Perspective of Sensorimotor Control
Status: Completed | Type: Observational
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: B-ER-109-188
Record Dates: First submitted 2021-06-20; First posted 2021-06-28 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Schizophrenia
Keywords: hand function; sensorimotor; motor control theory
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- schizophrenia group: No intervention age between 20-65, diagnosed schizophrenia by DSM-5.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention in this study

SUMMARY:
The study aims to explore the hand function in people with schizophrenia in the chronic stage.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20-65 years old
* Diagnosis with schizophrenia or schizoaffective disorder by psychiatrists according to DSM5.
* Remaining the same antipsychotics and the symptom was stable for at least one month before the study.
* Be able to follow comments and have sufficient cognitive ability assessed by Mini-Mental State Examination score >24

Exclusion Criteria:

* Substance abuse or other medical conditions that may affect movements.
* Using other non-antipsychotics that will affect movements in the same period.

Ages: 20 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants with schizophrenia will be recruited from the Department of Internal Medicine in National Cheng Kung University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2020-09-17 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Semmes Weinstein Monofilaments | baseline
  Semmes Weinstein Monofilaments is used to assess cutaneous pressure thresholds.
Pinch-holding-up-activity test | baseline
  The pinch apparatus is aims to assess the ability to modulate pinch force to movement-induced load fluctuations in a pinch-holding-up activity (PHUA).
Manual Tactile Test | baseline
  Manual tactile test (MTT) aims to assess the capacity of barognosis, roughness differentiation and stereognosis.
Purdue pegboard test | baseline
  The purpose for Purdue pegboard test is to measure manipulative dexterity including unimanual and bimanual hand dexterity.
The Valpar 8 simulates assembly work assessment | baseline
  Valpar8 simulates the light work and assess the ability of manual dexterity and motor coordination.

SECONDARY OUTCOMES:
Self-reported version of the graphic Personal and Social Performance (SRG-PSP) | baseline
  The self-reported version of the graphic personal and social performance is a self-report scale that aims to assess functional performance.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng-Kung University, Tainan, Taiwan

REFERENCES:
- [Derived] Lai YJ, Lin YC, Hsu CH, Tseng HH, Lee CN, Huang PC, Hsu HY, Kuo LC. Are the sensorimotor control capabilities of the hands the factors influencing hand function in people with schizophrenia? BMC Psychiatry. 2023 Nov 7;23(1):807. doi: 10.1186/s12888-023-05259-w. PMID 37936136